CLINICAL TRIAL: NCT01781000
Title: Training-induced Cerebral Reorganization in Schizophrenia
Brief Title: Cerebral Reorganization in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Prof. Dr. Brigitte Rockstroh, Prof. Dr., University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RO805/142
Record Dates: First submitted 2013-01-22; First posted 2013-01-31 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Schizophrenia
Keywords: Cognitive Training; Neuroplasticity; MEG; MATRICS
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Auditiory verbal discrimination training (Experimental): Brain Fitness & Brain Training- Posit Science
  Interventions: Behavioral: Brain Fitness & Brain Training- Posit Science
- Facial affect discrimination training (Experimental): Behavioral: Facial Affect Training- FAT
  Interventions: Behavioral: Facial Affect Training- FAT
- Treatment as usual (Active Comparator): standard treatment/rehabilitation protocol of schizophrenia ward
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Brain Fitness & Brain Training- Posit Science — Computer aided cognitive program designed for intensive training of auditory perception, memory and attention
  Arms: Auditiory verbal discrimination training
Behavioral: Facial Affect Training- FAT — Computer-aided cognitive program designed for intensive training of facial affect discrimination, memory and attention
  Arms: Facial affect discrimination training
Behavioral: Treatment as usual — standard treatment protocol of schizophrenia ward
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to reveal the specific effects of computer-aided cognitive training on cerebral reorganization in schizophrenia

DETAILED DESCRIPTION:
Impairment in cognitive functions is one of the main symptoms in schizophrenia and is currently one of the challenges in the treatment of the disease. In this study we compare effects of two computer-aided training programs. One focused on auditory perception and processing as a basic ability underlying higher order information processing. The other training focus on facial affect discrimination and working memory. Both trainings are computer-aided and time-intensive, including up to twenty sessions within four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia and disorders with psychotic features
* Intact auditory perception
* Intact visual perception

Exclusion Criteria:

* Mental retardation
* Age over 60
* Insufficient German language knowledge

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
change from baseline at post-intervention (4-weeks) and 3-months in each to the primary outcome measures: neuropsychological test scores (MCCB), MEG alpha oscillations | baseline, post-intervention (after 4 weeks), 3-months follow-up

SECONDARY OUTCOMES:
change from baseline in global functioning (GAF score) at 4 weeks and 3 months | baseline, post-intervention, 3-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Rockstroh, Prof. Dr., Study Chair — University Konstanz
Locations (1):
- University of Konstanz, Konstanz, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Popova P, Popov TG, Wienbruch C, Carolus AM, Miller GA, Rockstroh BS. Changing facial affect recognition in schizophrenia: effects of training on brain dynamics. Neuroimage Clin. 2014 Sep 4;6:156-65. doi: 10.1016/j.nicl.2014.08.026. eCollection 2014. PMID 25379427
- See also: Brain Training Software — http://www.positscience.com/